CLINICAL TRIAL: NCT07307768
Title: EEG Biomarker Development for Ketamine Administration
Brief Title: Ketamine Biomarker Validation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Soterix Medical (Industry)
Collaborators: Columbia University Irving Medical Center, New York, NY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KETAEEG
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression (TRD)
Keywords: Ketamine; EEG; Depression; MDD; unipolar Depression; Biomarker
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Depressive Disorder | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low level ketamine (Experimental): 0.25 mg/kg ketamine infusion
  Interventions: Drug: Ketamine (0.25 mg/kg)
- Medium level ketamine (Experimental): 0.5 mg/kg ketamine infusion
  Interventions: Drug: Ketamine (0.5 mg/kg)
- High level ketamine (Experimental): 0.75 mg/kg ketamine infusion
  Interventions: Drug: Ketamine (0.75 mg/kg)

INTERVENTIONS:
Drug: Ketamine (0.25 mg/kg) — Low level ketamine infusion therapy.
  Arms: Low level ketamine
Drug: Ketamine (0.5 mg/kg) — Medium level ketamine infusion therapy.
  Arms: Medium level ketamine
Drug: Ketamine (0.75 mg/kg) — High level ketamine infusion therapy.
  Arms: High level ketamine

SUMMARY:
We will be developing an EEG-based biomarker for the effects of ketamine infusion in patients with Depression. We will be analyzing the effects of ketamine infusion on Depression symptoms and EEG signals.

DETAILED DESCRIPTION:
This trial is a biomarker development study. We will be examining the effects of various doses of ketamine infusion on depressive symptoms and EEG signals in patients with unipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy patients who meet DMS-5 criteria for a major depressive episode (MDE) in the context of MDD and who score at least 22 on the Montgomery-Åsberg Depression Rating Scale (MADRS)
* If taking antidepressants, dose is stable for at least 6 weeks.

Exclusion Criteria:

* Lifetime history of bipolar disorder, schizoaffective disorder, schizophrenia, or any other psychotic disorder, including MDD with psychotic features
* A first-degree relative with bipolar disorder, schizoaffective disorder, or schizophrenia, with the potential participant younger than 33 years (i.e., still at age of risk for a psychotic disorder)
* Receipt of electroconvulsive therapy within 3 months of enrolling in the study
* History of IV drug use
* Nonresponse or intolerance to ketamine administered either clinically or as part of a prior research study
* Pregnancy, planning to conceive, or sexually active but not using adequate birth control.
* Actively suicidal (CSSRS≥3)
* No antipsychotics or medications (e.g. benzodiazepines, anti-epileptics) that are likely to interact with GABA or glutamate,

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) 22 | Baseline, Hour 1, Hour 4, Hour 24, and Hour 72
  Twenty-two question Depression rating scale (excluding the two questions on weight loss and diurnal variation)

SECONDARY OUTCOMES:
The Columbia Suicidality Severity Rating Scale (C-SSRS) | Baseline, Hour 1, Hour 4, Hour 24, and Hour 72
  A semi-structured, investigator-rated interview assessing both suicidal behavior and suicidal ideation.
The Clinician Administered Dissociative States Scale (CADSS) | Baseline, and Hour 1
  A scale that rates dissociative symptoms with a 27-item scale, rated 0-4, 19 subjective, and 8 observer items
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline and Hour 24
  A ten-item diagnostic used for the assessment of depression severity

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No